CLINICAL TRIAL: NCT01548521
Title: Tolerance of Intranasal Administration of OT in Prader-Willi Newborn Babies and Effect on Suck and Food Intake.
Brief Title: Tolerance of Intranasal Administration of OT in Prader-Willi Newborn Babies
Acronym: OTBB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10 152 02
Record Dates: First submitted 2011-12-30; First posted 2012-03-08 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi, neonates, poor suckling
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxytocin (Experimental)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 2 ui intranasal administration for the 3 first patients, 4UI for the 3 following patients.

SUMMARY:
Background: Prader-Willi syndrome (PWS) is a rare, complex multisystem genetic disorder arising from the lack of expression of paternally inherited imprinted genes on chromosome 15q11-q13. The syndrome includes severe neonatal hypotonia with impaired suckling leading to failure to thrive in the most severe cases, subsequently followed by an early onset of morbid obesity with insatiable hunger, combined with other endocrine dysfunction probably due to hypothalamic dysfunction. The pathophysiological mechanism of the occurrence of the 2 main nutritional phases of PWS is unknown. A deficit in the oxytocin (OT)-producing neurons of the paraventricular nucleus in the brain of these patients has been reported. In addition of its well-known anorexigenic effect, OT is involved in establishing and maintaining social codes. Indeed, we have recently shown in a double blind placebo study, that OT administration to adult patients with PWS significantly decreased depressive mood tendencies and tantrums while increasing trust in others with some data on a trend to decrease appetite with higher satiety. Moreover in a PWS mouse model generated from a MAGEL2 KO gene a single OT injection at 5 hr of life prevent the early death observed in 50 % of the new born mice by recovering normal suckling. Interestingly this effect is no longer observed if OT injection takes place later. These data, OT deficit in PWS, good tolerance of OT and its effect after intranasal administration in adult patients with PWS and the recent striking data obtained in the MAGEL2 mouse model, prompted us to evaluate the tolerance of a single administration of intranasal OT in PWS newborns and its possible effect on suckling and food intake. Nowadays the diagnosis of PWS is done during the first months of life in our country. At this age, children still present with poor suckling suggesting that OT may be still efficient. Moreover in adult patients with PWS we have shown that OT improves some typical behavioral troubles. Therefore we first want to evaluate the tolerance of the intranasal administration of OT in 6 infants with PWS genetically confirmed and its effect on suckling, milk intake and weight gain.

DETAILED DESCRIPTION:
We want to evaluate the tolerance of the intranasal administration of OT in 6 infants with PWS genetically confirmed and its effect on suckling, milk intake and weight gain. The three first patients will have single nasal administration of 2 IU of Oxytocin and, if no adverse event has been observed, the 3 following patients will have single nasal administration of 4 IU of Oxytocin. We will monitor cardiac pulse, blood pressure, urine emission and measure biological safety parameters (glycemia, natremia and kaliemia). Video will be performed during 1 day before the drug administration and the 3 days after in order to qualify the suckling. Quantitative evaluation of the milk intake during each feeding and per day will be also evaluated. Biological parameters will be measured OT, ghrelin, others neuroendocrine hormones involved in appetite regulation (leptin, cortisol, insulin, GLP-1, PYY, pancreatic polypeptide, orexin A, aMSH) taking advantage of blood samples for safety biological measurements. These infants will stay 8 days (which is less than the mean duration of hospitalization of these infants) with data records by phone at 1 month and then have a final visit after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* neonates with genetic diagnosis of Prader-Willi syndrome
* aged from 15 days to 5 months

Exclusion Criteria:

* exclusive tube feeding
* arrhythmia

Ages: 15 Days to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse event, description and quantification of their severity, imputability to oxytocin administration. | up to day 8

SECONDARY OUTCOMES:
Quantitative evaluation of food intake | from day 1 to month 3
  food intake is measured in ml
Evaluation of plasmatic OT, ghrelin and others neuroendocrine hormones involved in appetite regulation (leptin, cortisol, insulin, GLP-1, PYY, pancratic polypeptide, orexin A, aMSH) | from day 1 to month 3

CONTACTS AND LOCATIONS:
Overall Officials: Maithe TAUBER, MD, Principal Investigator — Hospital of Toulouse
Locations (1):
- Children Hospital of Toulouse Purpan, Toulouse, France